CLINICAL TRIAL: NCT04191824
Title: Genetic Testing to Understand and Address Renal Disease Disparities Across the United States
Acronym: GUARDD-US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH); Icahn School of Medicine at Mount Sinai (Other); University of Florida (Other); Indiana University School of Medicine (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00102997; U01HG010225 (NIH); U01HG007269 (NIH); U01HG010232 (NIH); U01HG010248 (NIH); U01HG010231 (NIH); U01HG010245 (NIH)
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease; Hypertension
Keywords: Kidney Disease; Genetic testing; APOL1; Genomics; Renal Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: Immediate versus delayed return of Apolipoprotein L1 (APOL1) genetic testing results to provider and participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Return of Results (Active Comparator): Immediate return of results to inform participant of APOL1 status (either positive or negative).
  Interventions: Other: Timing of return of results
- Delayed Return of Results (Active Comparator): Delayed return of results of APOL1 status (either positive or negative) after the completion of the 6 month final study visit.
  Interventions: Other: Timing of return of results

INTERVENTIONS:
Other: Timing of return of results — Participants will be randomized to immediate versus delayed APOL1 return of results

SUMMARY:
GUARDD-US is a prospective, multicenter, unblinded, two arm randomized pragmatic clinical trial. Participants will be randomized in a 1:1 ratio to immediate APOL1 gene testing and return of results (ROR) to participant and provider (Intervention arm) versus delayed APOL1 gene testing and ROR to participant and provider (Control arm). The main study will compare outcomes between APOL1 positive participants in the Intervention arm (i.e., early knowledge of APOL1 status) to APOL1 positive participants in the Control arm (i.e., delayed knowledge of APOL1 status). Participants that are APOL1 negative in the Intervention and Control groups will not be included in the main study analyses.

GUARDD-US also includes a substudy to determine the effect of knowledge of genetic test results that predict efficacy of various antihypertensive medications on change in SBP from baseline to 3 months in APOL1 negative individuals at participating sites.

This substudy is listed separately on clinicaltrials.gov as NCT06748040 and Unique Protocol ID - PRO00102997_A

DETAILED DESCRIPTION:
High-risk variants in the APOL1 gene explain approximately 70% of the excess prevalence of CKD in African Americans (AAs), conferring a 5 times higher risk for hypertensive CKD and a 10 times higher risk for ESRD. A pilot study (GUARDD), showed that returning APOL1 gene test results had a statistically significant improvement in SBP at 3 months when comparing APOL1 positives to APOL1 negatives who received their genetic testing results and when comparing APOL1 positives that received their results early to overall controls who did not receive their results until after the 3 month visit. GUARDD was not however powered to evaluate the effects of having and knowing a positive APOL1 status on outcomes for those with high risk of developing CKD (i.e., comparing outcomes for APOL1 positive patients who know their genetic risk to APOL1 positive patients who do not know their genetic risk). A broader trial is needed to better determine the importance of APOL1 gene testing for improving the testing, diagnosis, and treatment of individuals at risk of CKD.

The primary aim is to determine the effect of participant and provider knowledge of a positive APOL1 status and accompanying guideline based clinical decision support (CDS) on blood pressure management on change in systolic blood pressure (SBP) from baseline to 3 months after randomization among the APOL1 positive participants. Secondary aims are to:

1. Determine the effect of participant and provider knowledge of a positive APOL1 status on the probability of documented CKD diagnosis.
2. Determine the effect of participant and provider knowledge of a positive APOL1 status on the probability of receiving a urine microalbumin/creatinine testing and ACE-I/ARB prescription based on results of the urine microalbumin level.
3. Explore cost effectiveness, mediators, moderators, psychobehavioral impact of results disclosure on participants, and effects of participant and provider knowledge of APOL1 status on provider treatment recommendations.

Approximately 6,750 participants of African ancestry age 18-70 with hypertension that either: 1) do not have diabetes and do not have CKD, or 2) have CKD. Participants with diabetes may be included as long as they also have CKD.

Population for Main Study:

Participants from Randomized Population (above) who test positive for APOL1

Main Study Analyses:

* To determine the effect of participant and provider knowledge of a positive APOL1 status on SBP, we will compare the change in SBP from baseline to 3 months of the Intervention - APOL1 positive group to the change in SBP from baseline to 3 months of the Control - APOL1 positive group using a two sided t-test, as appropriate, with an overall two-sided type I error of 0.05.
* The effect of knowledge of a positive APOL1 status on all secondary endpoints will be compared between Intervention - APOL1 positives to Control - APOL1 positives with the proportion difference test.
* Additional analyses will include analysis of time trends in SBP, subset analyses, and exploratory analyses of cost effectiveness, mediators, moderators, psychobehavioral impact of results disclosure on participants, and effects of knowledge of APOL1 status on provider treatment recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Self reported African ancestry
* English Speaking
* Age 18-70 years
* Have diagnosis of hypertension: Diagnosis of hypertension is defined by either:

  * ICD10 diagnosis codes (i.e., I10; I11.x; I12.x; I13.x; I16.x) OR
  * On active antihypertensive therapy for indication of hypertension OR
  * Having systolic blood pressure of 140 mm Hg or greater in at least 2 of the last 3 consecutive recorded values in the EHR OR
  * Having hypertension in the patient's medical record problem list
* Have been seen at ≥1 time in past year at a participating primary care site
* Either: 1) do not have diabetes and do not have CKD, or 2) have CKD; Participants with diabetes may be included as long as they also have CKD.

CKD is defined by either: A) ICD10 codes (i.e., N18.x; E08.22; E09.22; E10.22; E11.22;E13.22 (exclude Z94.0; N18.6; Z99.2)) OR B) Microalbumin/proteinuria level >30 mg/g for 2 time periods ≥ 3 months. Values taken within 12 months of enrollment, unless 2 values are unavailable, then review within 24 months of enrollment. OR C) 15 ≤ eGFR ≤ 60 ml/min for 2 time periods ≥ 3 months. GFRs are taken within 12 months of enrollment, unless 2 values are unavailable, then review within 24 months.

Diabetes is defined by: HbA1c ≥ 6.5 at least one time in the last year OR ICD10 diagnosis codes OR Having diabetes in the patient's medical record problem list.

Exclusion Criteria:

* Have diabetes, but no CKD.
* Are currently on dialysis (ICD 10 codes N18.6, Z99.2 and Z94.0)
* Have ESRD (eGFR<15 ml/min)
* Have a left ventricular assist device (LVAD)
* Have a terminal illness
* Have patient-reported known pregnancy at time of enrollment
* Have had a liver, kidney, or allogeneic bone marrow transplant
* Too cognitively impaired to provide informed consent and/or complete the study protocol
* Institutionalized or too ill to participate (i.e. incarcerated, psychiatric or nursing home facility)
* Plan to move out of the area within 6 months of enrollment
* Not a current patient seeing a provider who cares for their hypertension (i.e., family medicine, internal medicine, nephrology, HIV provider, cardiology, hypertension specialists) at a participating site
* Previously participated in the GUARDD pilot study OR have previously undergone APOL1 testing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6789 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hrishikesh Chakraborty, DrPH, Study Director — Duke University; Carol Horowitz, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida - Gainesville, Gainesville, Florida
  - University of Florida - Jacksonville, Jacksonville, Florida
  - Eskenazi Health, Indianapolis, Indiana
  - Indiana University, Indianapolis, Indiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Institute for Family Health, New York, New York
  - Southeastern Healthcare, Lumberton, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Meharry Medical College, Nashville, Tennessee
  - Nashville General Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
The Data Coordinating Center (DCC) will submit de-identified participant level datasets and associated documentation to the NHGRI's data repository - Genomic Analysis, Visualization and Informatics Lab-space (AnVIL), for use by other investigators. The datasets and associated documentation will be available after publication of the primary results manuscript. Documentation will include annotated case report forms, list of derived variables along with descriptions, and a description of the data model and de-identification process.
Supporting Information: Study Protocol, ICF
Time Frame: 3 months after publication
Access Criteria: Datasets will be designated as controlled access and researchers will be able to apply to NIH data access committees (DACs) for use of these datasets.

REFERENCES:
- [Background] Eadon MT, Cavanaugh KL, Orlando LA, Christian D, Chakraborty H, Steen-Burrell KA, Merrill P, Seo J, Hauser D, Singh R, Beasley CM, Fuloria J, Kitzman H, Parker AS, Ramos M, Ong HH, Elwood EN, Lynch SE, Clermont S, Cicali EJ, Starostik P, Pratt VM, Nguyen KA, Rosenman MB, Calman NS, Robinson M, Nadkarni GN, Madden EB, Kucher N, Volpi S, Dexter PR, Skaar TC, Johnson JA, Cooper-DeHoff RM, Horowitz CR; GUARDD-US Investigators. Design and rationale of GUARDD-US: A pragmatic, randomized trial of genetic testing for APOL1 and pharmacogenomic predictors of antihypertensive efficacy in patients with hypertension. Contemp Clin Trials. 2022 Aug;119:106813. doi: 10.1016/j.cct.2022.106813. Epub 2022 Jun 1. PMID 35660539

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by providers who care for participants with hypertension (including, for example, general internists, primary care providers, and nephrologists).
Pre-assignment Details: There were 6789 participants consented into the overall GUARDD-US trial. Of the 6789, 35 consented participants were not randomized into the trial and were not assigned to a treatment arm. The remaining 6754 consented participants were randomized and assigned into the treatment arms. The 6754 randomized participants will be described moving forward.
Period: Overall Study
Arm/Group | Immediate Return of Results | Delayed Return of Results
Started | 3380 | 3374
Completed | 2869 | 2884
Not Completed | 511 | 490
Not completed — Death | 13 | 12
Not completed — Lost to Follow-up | 456 | 435
Not completed — Physician Decision | 2 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 16 | 18
Not completed — Early site closure | 24 | 22

BASELINE CHARACTERISTICS:
Population: ITT refers to the Intent To Treat population, while mITT, a subset of ITT, refers to the modified Intent To Treat population. The mITT population is the primary analytical population, consisting of ITT participants with APOL1 positive phenotype. APOL1 positive phenotype refers to participants with 2 high risk alleles at the APOL1 locus (APOL1-HR).
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Return of Results | Delayed Return of Results | Total
Number analyzed (Participants) | 3380 | 3374 | 6754
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Intent to Treat population
  years | 55.3 (10.3) | 55.4 (10.2) | 55.3 (10.3)
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Modified Intent to Treat population
  years
    number analyzed (Participants) | 486 | 468 | 954
    (all) | 54.7 (9.9) | 55.1 (10.1) | 54.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Intent to Treat population. Data not collected on one Delayed Return of Results participant.
  Participants
    number analyzed (Participants) | 3380 | 3373 | 6753
    Female | 2178 | 2132 | 4310
    Male | 1202 | 1241 | 2443
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Modified Intent to Treat population
  Participants
    number analyzed (Participants) | 486 | 468 | 954
    Female | 326 | 274 | 600
    Male | 160 | 194 | 354
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Intent to Treat population
  Participants
    Hispanic or Latino | 79 | 95 | 174
    Not Hispanic or Latino | 3281 | 3258 | 6539
    Unknown or Not Reported | 20 | 21 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Modified Intent to Treat population
  Participants
    number analyzed (Participants) | 486 | 468 | 954
    Hispanic or Latino | 3 | 8 | 11
    Not Hispanic or Latino | 478 | 457 | 935
    Unknown or Not Reported | 5 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Intent to Treat population
  Participants
    Race: American Indian or Alaska Native | 10 | 9 | 19
    Race: Asian | 1 | 0 | 1
    Race: Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
    Race: Black or African American | 3101 | 3090 | 6191
    Race: White | 0 | 1 | 1
    Race: North African/Mediterranean | 2 | 0 | 2
    Race: More than one race | 184 | 190 | 374
    Race: Unknown or Not Reported | 79 | 83 | 162
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Modified Intent to Treat population
  Participants
    Race: number analyzed (Participants) | 486 | 468 | 954
    Race: American Indian or Alaska Native | 0 | 2 | 2
    Race: Asian | 0 | 0 | 0
    Race: Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
    Race: Black or African American | 457 | 428 | 885
    Race: White | 0 | 0 | 0
    Race: North African/Mediterranean | 1 | 0 | 1
    Race: More than one race | 17 | 28 | 45
    Race: Unknown or Not Reported | 10 | 9 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3380 | 3374 | 6754

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure From Baseline to 3 Months for APOL1 Positive Participants.
Time Frame: Baseline to 3 month study visit
Population: Modified Intent To Treat (mITT) population, consisting of ITT participants with APOL1 positive phenotype (APOL1-HR).
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Immediate Return of Results (Modified Intent to Treat, mITT): Immediate return of results to APOL1 positive participants.
- Delayed Return of Results (Modified Intent to Treat, mITT): Delayed return of results to APOL1 positive participants after the completion of the 6 month final study visit.
Arm/Group | Immediate Return of Results (Modified Intent to Treat, mITT) | Delayed Return of Results (Modified Intent to Treat, mITT)
Number analyzed (Participants) | 446 | 428
mmHg | -1.8 (18.8) | -1.5 (17.3)
Statistical Analysis 1: Comparison: Immediate Return of Results (Modified Intent to Treat, mITT) vs Delayed Return of Results (Modified Intent to Treat, mITT); Test type: Superiority; p = 0.7769, t-test, 2 sided — In order to maintain an overall alpha of 0.05 and account for two interim analyses, a two-sided alpha of 0.0492 was used for assessing the statistical significance in the final analysis of this primary endpoint; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-2.7 to 2.1]

2. Secondary Outcome: Change in Number of Participants With Urine Microalbuminuria/Proteinuria Orders
Time Frame: Baseline to 6 month study visit
Population: Modified Intent To Treat (mITT) population, consisting of ITT participants with APOL1 positive phenotype (APOL1-HR).
Measure: Count of Participants; unit: Participants
Groups:
- Immediate Return of Results (Modified Intent to Treat, mITT): Immediate return of results to APOL1 positive participants (APOL1-HR).
- Delayed Return of Results (Modified Intent to Treat, mITT): Delayed return of results to APOL1 positive participants (APOL1-HR) after the completion of the 6 month final study visit.
Arm/Group | Immediate Return of Results (Modified Intent to Treat, mITT) | Delayed Return of Results (Modified Intent to Treat, mITT)
Number analyzed (Participants) | 473 | 454
Participants | 95 | 43
Statistical Analysis 1: Comparison: Immediate Return of Results (Modified Intent to Treat, mITT) vs Delayed Return of Results (Modified Intent to Treat, mITT); Test type: Superiority; p < 0.0001, Chi-squared; Risk Difference (RD) = 0.106, 95% CI 2-sided [0.061 to 0.151]

3. Secondary Outcome: Number of Participants With Documented Order of Microalbuminuria/Proteinuria Tests
Time Frame: From baseline to 6 month study visit
Population: Modified Intent To Treat (mITT) population, consisting of ITT participants with APOL1 positive phenotype (APOL1-HR).
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Return of Results (Modified Intent to Treat, mITT) | Delayed Return of Results (Modified Intent to Treat, mITT)
Number analyzed (Participants) | 473 | 454
Participants | 302 | 264
Statistical Analysis 1: Comparison: Immediate Return of Results (Modified Intent to Treat, mITT) vs Delayed Return of Results (Modified Intent to Treat, mITT); Test type: Superiority; p = 0.0753, Chi-squared; Risk Difference (RD) = 0.057, 95% CI 2-sided [-0.006 to 0.120]

4. Secondary Outcome: Number of Participants With a Change in Documented Diagnosis for Stage 3 CKD and Above
Time Frame: From baseline to 6 month study visit
Population: Modified Intent To Treat (mITT) population, consisting of ITT participants with APOL1 positive phenotype (APOL1-HR).
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Return of Results (Modified Intent to Treat, mITT) | Delayed Return of Results (Modified Intent to Treat, mITT)
Number analyzed (Participants) | 456 | 441
Participants | 6 | 5
Statistical Analysis 1: Comparison: Immediate Return of Results (Modified Intent to Treat, mITT) vs Delayed Return of Results (Modified Intent to Treat, mITT); Test type: Superiority; p = 0.8044, Chi-squared; Risk Difference (RD) = 0.002, 95% CI 2-sided [-0.013 to 0.016]

5. Secondary Outcome: Number of Participants With Documented Diagnosis of CKD Stage 3 and Above
Time Frame: From baseline to 6 month study visit
Population: Modified Intent To Treat (mITT) population, consisting of ITT participants with APOL1 positive phenotype (APOL1-HR).
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Return of Results (Modified Intent to Treat, mITT) | Delayed Return of Results (Modified Intent to Treat, mITT)
Number analyzed (Participants) | 456 | 441
Participants | 83 | 103
Statistical Analysis 1: Comparison: Immediate Return of Results (Modified Intent to Treat, mITT) vs Delayed Return of Results (Modified Intent to Treat, mITT); Test type: Superiority; p = 0.0570, Chi-squared; Risk Difference (RD) = -0.052, 95% CI 2-sided [-0.105 to 0.002]

6. Secondary Outcome: Number of Participants With a Change in Documented Diagnosis for Any Stage CKD
Time Frame: From baseline to 6 month study visit
Population: Modified Intent To Treat (mITT) population, consisting of ITT participants with APOL1 positive phenotype (APOL1-HR).
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Return of Results (Modified Intent to Treat, mITT) | Delayed Return of Results (Modified Intent to Treat, mITT)
Number analyzed (Participants) | 456 | 441
Participants | 31 | 10
Statistical Analysis 1: Comparison: Immediate Return of Results (Modified Intent to Treat, mITT) vs Delayed Return of Results (Modified Intent to Treat, mITT); Test type: Superiority; p = 0.0012, Chi-squared; Risk Difference (RD) = 0.045, 95% CI 2-sided [0.018 to 0.072]

7. Secondary Outcome: Number of Participants With Documented Diagnosis of All Stages of CKD
Time Frame: From baseline to 6 month study visit
Population: Modified Intent To Treat (mITT) population, consisting of ITT participants with APOL1 positive phenotype (APOL1-HR).
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Return of Results (Modified Intent to Treat, mITT) | Delayed Return of Results (Modified Intent to Treat, mITT)
Number analyzed (Participants) | 456 | 441
Participants | 140 | 138
Statistical Analysis 1: Comparison: Immediate Return of Results (Modified Intent to Treat, mITT) vs Delayed Return of Results (Modified Intent to Treat, mITT); Test type: Superiority; p = 0.8483, Chi-squared; Risk Difference (RD) = -0.006, 95% CI 2-sided [-0.066 to 0.055]

ADVERSE EVENTS:
Time Frame: 6 months
Description: GUARDD-US does not include a drug or device intervention. For this reason, no adverse events (other than all-cause mortality) were collected or recorded in the study database.
Groups:
- Immediate Return of Results (Intent to Treat, ITT): Immediate return of results to inform participant of APOL1 status (either positive or negative).
- Delayed Return of Results (Intent to Treat, ITT): Delayed return of results of APOL1 status (either positive or negative) after the completion of the 6 month final study visit.
Arm/Group | Immediate Return of Results (Intent to Treat, ITT) | Delayed Return of Results (Intent to Treat, ITT)
All-Cause Mortality (participants affected / at risk) | 13/3380 | 12/3374
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT04191824/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT04191824/ICF_000.pdf